CLINICAL TRIAL: NCT02330601
Title: Effect of Endoscopic Papillary Large Balloon Dilation on Recurrent Rate of Patients With Recurrentstones in Bile Duct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20140424-6
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Endoscopic Papillary Large Balloon Dilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): The papilla orifice could be enlarged by asphincterotomeif necessary. The stones were retrieved by a basket or a retrieval balloon
- EPLBD group (Other): a CRE balloon (diameter 10, 11, 12, 13.5, 15 mm; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast. When the waist disappeared, the balloon was kept inflated for 120s. The stones were then retrieved by a basket or a retrieval balloon.Mechanical lithotripsy was used if necessary
  Interventions: Procedure: endoscopic papillary large balloon dilation

INTERVENTIONS:
Procedure: endoscopic papillary large balloon dilation — For the patients in EPLBD group, a CRE balloon (diameter 10, 11, 12, 13.5, 15 mm; Boston Scientific) was chosen according to the diameter of bile duct. It was placed across the papilla orifice and then gradually filled with diluted contrast. When the waist disappeared, the balloon was kept inflated for 120s. The stones were then retrieved by a basket or a retrieval balloon.Mechanical lithotripsy was used if necessary
  Other Names: EPLBD
  Arms: EPLBD group

SUMMARY:
The recurrent rate of CBDS in patients with recurrent CBDS is high. It was reported that up to 60% of patients had stone recurrence within two years after stone retrieval by ERCP. Although EPLBD is useful for for extraction of large CBDS with less operation time and mechanical lithotripsy.It is not known whether EPLBD could prevent the recurrence in patients with recurrent CBDS.Although Harada et al found that EPLBD might reduce the short-term recurrence of CBD stones in patients with previous ES. It is a retrospective study with a small sample size (n=94).

Here a prospective, randomized controlled study including two tertiary centers was designed. The aim of this study was to investigate whether EPLBD could reduce the recurrence rate in patients with recurrent CBDS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Patients with recurrent CBDS after ERCP

Exclusion Criteria:

1. Benign or malignant CBD stricture
2. Recurrent stone within 3 months after ERCP
3. Previous endoscopic papillary large balloon dilation (EPLBD)
4. Prior surgery of Bismuth II and Roux-en-Y
5. Septic shock
6. Coagulopathy (INR>1.3), platelet<50000 or using anti-coagulation drugs
7. With expected life span less than 24 months
8. Pregnant women
9. Refusal or unable to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Recurrent rate of CBDS within two years after ERCP | up to 2 years
  Within the two years after ERCP, CBDS was found again by CT, MRCP, ERCP or biliary surgery

SECONDARY OUTCOMES:
recurrent time | up to 2 years
success rate of stone extraction | up to 2 years
success rate of stone extraction in the initial attempt | up to 2 years
performance time of ERCP | up to 2 years
rate of mechanical lithotripsy | up to 2 years
post-ERCP complication | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Xijing Hospital of Digestive Diseases.The Fourth Military Medical University
Locations (2):
- China (2):
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi

REFERENCES:
- [Background] Yoon HG, Moon JH, Choi HJ, Kim DC, Kang MS, Lee TH, Cha SW, Cho YD, Park SH, Kim SJ. Endoscopic papillary large balloon dilation for the management of recurrent difficult bile duct stones after previous endoscopic sphincterotomy. Dig Endosc. 2014 Mar;26(2):259-63. doi: 10.1111/den.12102. Epub 2013 Apr 14. PMID 23581623
- [Result] Stefanidis G, Viazis N, Pleskow D, Manolakopoulos S, Theocharis L, Christodoulou C, Kotsikoros N, Giannousis J, Sgouros S, Rodias M, Katsikani A, Chuttani R. Large balloon dilation vs. mechanical lithotripsy for the management of large bile duct stones: a prospective randomized study. Am J Gastroenterol. 2011 Feb;106(2):278-85. doi: 10.1038/ajg.2010.421. Epub 2010 Nov 2. PMID 21045816
- [Derived] Wang X, Wang X, Sun H, Ren G, Wang B, Liang S, Zhang L, Kang X, Tao Q, Guo X, Luo H, Pan Y. Endoscopic Papillary Large Balloon Dilation Reduces Further Recurrence in Patients With Recurrent Common Bile Duct Stones: A Randomized Controlled Trial. Am J Gastroenterol. 2022 May 1;117(5):740-747. doi: 10.14309/ajg.0000000000001690. Epub 2022 Feb 16. PMID 35191430